CLINICAL TRIAL: NCT05145673
Title: Effect of Aqueous Cinnamon Extract on the Postprandial Glycaemia Levels in Type 2 Diabetes Mellitus: a Randomized Controlled Trial
Brief Title: Effect of Aqueous Cinnamon Extract on the Postprandial Glycaemia Levels in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 525cinnamon
Record Dates: First submitted 2021-11-10; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (OGTT) (Placebo Comparator): The control group was given an glucose solution to oral glucose tolerance test (OGTT) .
  Interventions: Other: Placebo (OGTT)
- Cinnamon (OGTT plus aqueous cinnamon extract) (Experimental): The Experimental group was given an glucose solution to oral glucose tolerance test (OGTT) followed by aqueous cinnamon extract.
  Interventions: Other: Cinnamon (OGTT plus aqueous cinnamon extract)

INTERVENTIONS:
Other: Placebo (OGTT) — The control group was given an glucose solution to oral glucose tolerance test (OGTT) The glucose solution consist in a glucose drink with 75g of anhydrous D-Glucose dissolved in 200 mL of water at room temperature, as prescribed by ADA. The blood glucose levels were measured before intervention at fasting (t0) and after 30 (t30), 60 (t60, 90 (t90) and 120 (t120) minutes after intervention from both groups.
  Arms: Placebo (OGTT)
Other: Cinnamon (OGTT plus aqueous cinnamon extract) — The intervention group was given an glucose solution to OGTT followed by a cinnamon aqueous extract. The glucose solution consist in a glucose drink with 75g of anhydrous D-Glucose dissolved in 200 mL of water at room temperature, as prescribed by ADA. The blood glucose levels were measured before intervention at fasting (t0) and after 30 (t30), 60 (t60, 90 (t90) and 120 (t120) minutes after intervention from both groups.
  Arms: Cinnamon (OGTT plus aqueous cinnamon extract)

SUMMARY:
The type 2 diabetes mellitus is a chronic disease and it is a highly prevalent globally. Cinnamon is a spicy used on the traditional cuisine, which have as been associated with beneficial effects on postprandial blood glucose levels (BGL). The aim of the present study was to investigate the effect of cinnamon tea (6g C. burmannii/100mL) on postprandial glycaemia in type 2 diabetic adults.

Following ethical committee approval, thirty-six subjects were selected and randomly allocated in 2 groups (n=18): cinnamon group, which was administrated OGTT (oral glucose tolerance test) followed by cinnamon tea; control group, which was administrated only OGTT. At baseline, anthropometric data, medical condition and pharmacological therapy were collected. A 24-hour dietary recall was taken preceding each intervention. Food Processor SQL (version 10.5.9) program was used to analyze the food nutritional composition. Chemical analysis was performed for total phenols determinations (adapted from Prabha et al) and antioxidant activity for FRAP and for DPPH tests (adapted from K. Thaipong et al.) Statistical analysis was performed using SPSS Statistics program. Data are mean±SEM.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (DM2) subjects aged between 35-77 years were recruited into this study through nutrition appointment, Holon Pharmacy from Lisbon and Portalegre, Portugal. After the approval of the Ethics Committee, 36 individuals, were selected and invited to participate in this study. After eligibility criteria applied, a randomized controlled clinical trial, blind to participants, was conducted to 36 DM2 subjects. Participants were randomly assigned to intervention (n=18) or control group (n=18). The first participant of the study was randomly allocated to intervention or control group and the following participants were systematically allocated in each group. The anonymity and the confidentiality of the participants data collected were guaranteed through a code attributed to each participant. The control group was given a glucose solution to oral glucose tolerance test (OGTT) and the intervention group was given a glucose solution to OGTT followed by a cinnamon aqueous extract. The glucose solution consist in a glucose drink with 75g of anhydrous D-Glucose dissolved in 200 mL of water at room temperature, as prescribed by ADA. The blood glucose levels were measured before intervention at fasting (t0) and after 30 (t30), 60 (t60, 90 (t90) and 120 (t120) minutes after intervention from both groups.

Aqueous cinnamon extract was prepared by Cinnamomum burmannii bark (from Sucrame Company, Portugal) with Indonesia origin. Sticks of cinnamon (60 g) were soaked into 1000 mL of water. After 24 h at room temperature, cinnamon solution was heated for 30 min at 100°C and then filtered at room temperature. After the cinnamon tea preparation a 100 mL individual dose was distributed to each participant. For chemical analysis, a hydromethanolic extract (50 : 50) was performed with aqueous cinnamon extract previously obtained.

Anthropometric paraments and pharmacological therapy data were collected at the beginning of the study. At day before the intervention, a 24-hour food recall questionnaire was employed to participants of the study and carefully instructed by an investigator to complete the food record. The Food Processor SQL (10.14.2. version) programme was applied to analysed the nutritional composition of meals, such as, total energy intake (Kcal), proteins (g), lipids (g), carbohydrates (g), dietary fibre (g) and soluble fibre (g). It were also estimated the glycemic index and glycemic load of food intake.

Based on the blood glucose values, the blood glucose incremental area under the curve (AUCi) of each participant was defined using the GraphPad Prism program (version 5.0). Maximum concentrations (Cmax) and variations of maximum concentrations (ΔCmax) were determined by comparing with its respective baseline glycemia levels values.

The total phenolic concentration in the C. burmanni extract was determined according to Folin-Ciocalteu method employing gallic acid as standard. For the determination of antioxidant activity two methods were performed: FRAP and DPPH, adapted by Thaipong et al. The FRAP method for determination of ferric reducing effect was based on the reduction, at low pH, employing a colourless ferric complex (Fe3+) to a blue-coloured ferrous complex (Fe2+) by electron-donating antioxidants action in 2,4,6-tri(2-pyridyl)-s-triazine (TPTZ) presence.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 18 years or older
* subjects with DM2 diagnostic and men or non-pregnant women.

Exclusion Criteria:

* insulin-treated subjects
* history of gastrointestinal symptoms/diseases
* allergy to cinnamon
* fasting less than 8 hours
* cinnamon intake at day before the intervention
* intense exercise until 2 hours before the intervention

Ages: 35 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose levels at beginning | At beginning (before intervention)
  Mean values of blood glucose levels from both control and experimental groups
Blood glucose levels at 30 minutes | At 30 minutes after intervention
  Mean values of blood glucose levels from both control and experimental groups
Blood glucose levels at 60 minutes | At 60 minutes after intervention
  Mean values of blood glucose levels from both control and experimental groups
Blood glucose levels at 90 minutes | At 90 minutes after intervention
  Mean values of blood glucose levels from both control and experimental groups
Blood glucose levels at 120 minutes | At 120 minutes after intervention
  Mean values of blood glucose levels from both control and experimental groups
Incremental area under the curve of blood glucose | At 120 minutes after intervention
  Based on the blood glucose values, the blood glucose incremental area under the curve (AUCi) of each participant was defined using the GraphPad Prism program (version 5.0)
Variation of blood glucose maximum concentration | At 60 minutes after intervention
  Mean values of glucose maximum concentration variation

SECONDARY OUTCOMES:
Anthropometric parameters - body weight | At baseline
  Mean values of body weight (in kilogram - Kg)
Anthropometric parameters - height | At baseline
  Mean values of Height (in centimeters - cm)
Anthropometric parameters - waist circumference | At baseline
  Mean values of waist circumference (in centimeters - cm)
Anthropometric parameters - body mass index | At baseline
  Mean values of body mass index (Kg/m2), calculated as weight (Kg) divided by height (m2) squared (Kg/m2)
Anthropometric parameters - Skeletal muscle mass | At baseline
  Mean values of Skeletal muscle mass (in kilogram - Kg)
Anthropometric parameters - visceral fat | At baseline
  Mean values of visceral fat (cm3)
Pharmacological therapy | At baseline
  Percentage of antidiabetic orals (biguanide, sulfonylurea, alpha-glucosidase inhibitor, dipeptidyl peptidase 4 inhibitors
Total protein intake | At baseline
  Means values of total protein intake (in grams - g) obtained through The Food Processor SQL software
Total lipid intake | At baseline
  Means values of total lipid intake (in grams - g) obtained through The Food Processor SQL software
Total carbohydrate intake | At baseline
  Means values of total carbohydrate intake (in grams - g) obtained through The Food Processor SQL software
Total energy intake | At baseline
  Means values of total energy intake (in kilocalorie - Kcal) obtained through The Food Processor SQL software
Total polyphenols content | At baseline
  Mean values of total polyphenols content of cinnamon extract (mg/L equivalent of gallic acid)
Antioxidant activity | At baseline
  Mean values of antioxidant activity of cinnamon extract by FRAP and DPPH assays (micromol Trolox/L)